CLINICAL TRIAL: NCT03532243
Title: Acute Effects of Incremental Inspiratory Loads on Respiratory Mechanics and Neural Respiratory Drive(NRD) in Patient With Stable Chronic Obstructive Pulmonary Disease(COPD).
Brief Title: Acute Effects of Incremental Inspiratory Loads on Respiratory Mechanics and NRD in Patient With Stable COPD.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-HXNK-007
Record Dates: First submitted 2018-03-26; First posted 2018-05-22 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2018-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; inspiratory muscle training; Central Drive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- respiratory muscle weakness (Experimental): Patients with respiratory muscle weakness are performing the threshold loading device with incremental inspiratory load.
  Interventions: Procedure: incremental inspiratory load
- normal respiratory muscle (Experimental): Patients with normal respiratory muscle are performing the threshold loading device with incremental inspiratory load.
  Interventions: Procedure: incremental inspiratory load

INTERVENTIONS:
Procedure: incremental inspiratory load — inspiratory load ranges between 10 and 40 cm water column (cmH2O)or intolerable to the patient, each load increment for 5cm water column.

SUMMARY:
Inspiratory muscle training has been an important part of pulmonary rehabilitation program directed at patients with COPD. It can increase respiratory muscle strength, relieve dyspnea ,improve the quality of life in COPD patients. However, there is no uniform standard for the intensity of inspiratory muscle training. By comparing a series of indexes, such as maximal inspiratory pressure, maximal expiratory pressure, degree of dyspnea and exercise capacity before and after the training under different intensity, a large number of literatures have explored the appropriate intensity of inspiratory muscle training. But to date, there are few studies about the effects of different intensity of inspiratory muscle training on respiratory physiological mechanism. It has been shown that inspiratory muscle training may be more beneficial to improve the pulmonary rehabilitation effect of COPD patients with inspiratory muscle weakness. So it is not clear whether there is a difference in respiratory physiology between patients with normal inspiratory muscle strength and those with lower inspiratory muscle strength. Respiratory central drive, as an important physiological index, which can be reflected by minute ventilation volume, mouth pressure, mean inspiratory flow and diaphragm electromyography,is closely related to the symptoms and the severity of the disease.Therefore,the purpose of this study was to investigate the changes of respiratory mechanics and central drive in COPD patients at different inspiratory loads, and at the same loads between patients with and without respiratory muscle weakness.That can provide more evidential evidence for setting up the intensity of inspiratory muscle training.

DETAILED DESCRIPTION:
The patients with COPD will be admitted in one intervention groups(performing on threshold loading device).Before using threshold loading device, we will measure the relevant parameters of lung volume, respiratory flow,diaphragm electromyogram, central drive mechanical and other baseline index.Then incremental inspiratory load will be applied to investigate the effects of inspiratory load on the above mentioned respiratory mechanics parameters.

ELIGIBILITY:
Inclusion Criteria:

- Patients with pulmonary function test of forced expiratory volume at one second (FEV1)/forced vital capacity(FVC) < 70% after inhalation of bronchial dilation agent. Patients in a clinically stable state.

Exclusion Criteria:

- Patients were excluded if they had other respiratory diseases ,or evidence of pneumothorax or mediastinal emphysema and pacemaker installed.

Patients with acute cardiovascular event and severe cor pulmonale. Patients with poor compliance. An Other causes of diaphragmatic dysfunction

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Diaphragmatic function | Change from baseline in diaphragm electromyogram at the load of 10cm water column (cmH2O).(1 minutes later,3 minutes later,5 minutes later,7 minutes later,9 minutes later,11 minutes later, 13 minutes later)
  Diaphragmatic function can be assessed by diaphragm electromyogram (EMGdi), which reflect the physiological activity of the diaphragm and indicate functional status of the central drive.

SECONDARY OUTCOMES:
Respiratory pressure | Change from baseline in respiratory pressure at the load of 10cm water column (cmH2O).(1 minutes later,3 minutes later,5 minutes later,7 minutes later,9 minutes later,11 minutes later, 13 minutes later)
  Respiratory pressure can be assessed by transdiaphragmatic pressure ( Pdi).
Respiratory volume | Change from baseline in respiratory volume at the load of 10cm water column (cmH2O).(1 minutes later,3 minutes later,5 minutes later,7 minutes later,9 minutes later,11 minutes later, 13 minutes later)
  Respiratory volume can be assessed by Tidal volume (VT).
Degree of dyspnea | Change from baseline in degree of dyspnea at the load of 10cm water column (cmH2O).(1 minutes later,3 minutes later,5 minutes later,7 minutes later,9 minutes later,11 minutes later, 13 minutes later)
  Difference in the degree of dyspnea can be measured by Borg index.

OTHER OUTCOMES:
Pulse oxygen saturation (SpO2) | Change from baseline in pulse oxygen saturation at the load of 10cm water column (cmH2O).(1 minutes later,3 minutes later,5 minutes later,7 minutes later,9 minutes later,11 minutes later, 13 minutes later)
  Change in SpO2 can be recorded by noninvasive monitoring instruments.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Chen, Doctor, Principal Investigator — Zhujiang Hospital,Southern Medical Unversity
Locations (1):
- Zhujiang Hospital,Southern Medical Universtiy, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No